CLINICAL TRIAL: NCT03455192
Title: The Effect of Synbiotic Tablet Usage on the Clinical and Biochemical Parameters in Smokers and Nonsmokers With Gingivitis: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Synbiotic as an Adjunct to Mechanical Treatment of Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Nuray Ercan, Principal Investigator, Kırıkkale University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/01
Record Dates: First submitted 2018-02-16; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Gingivitis; Chronic; Smoking
Keywords: gingivitis; gingival crevicular fluid; probiotics; smoking; periodontal medicine
MeSH Terms: conditions — Gingivitis; Bronchiolitis Obliterans Syndrome; Smoking

STUDY DESIGN:
Intervention Model Description: double-blind randomized placebo-controlled clinical trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic supplements (Experimental): One synbiotic tablet, per day, during 30 days
  Interventions: Drug: Synbiotic Supplement
- Placebo Oral Tablet (Placebo Comparator): One placebo tablet , per day, during 30 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Synbiotic Supplement
  Other Names: NOBEL (NBL) Probiotic Optima
  Arms: Synbiotic supplements
Drug: Placebo Oral Tablet
  Arms: Placebo Oral Tablet

SUMMARY:
The aim of this study is to evaluate the efficacy of oral administration of synbiotic tablets on the clinical parameters and the levels of selected inflammatory mediators in gingival crevicular fluid (GCF) in smokers and non-smokers with gingivitis.

This study designed as a double-blind randomized placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Some patients like smokers have ongoing host response even after bacterial plaque removal achieved. Therefore efforts to develop effective treatment approaches remain an important objective in the treatment of gingivitis to prevent periodontitis especially in patients at high risk for developing periodontitis as smokers.

Smoking is a major risk factor for the incidence and the progression of periodontal diseases. The increased periodontal disease susceptibility in smokers is predominantly caused by changes in inflammatory and immune responses. Cigarette smoking also influences the amount and the composition of subgingival plaque. Smokers have higher numbers of pathogens in their resident biofilm and display an ongoing host response even after biofilm removal. Different approaches were explored to reduce the negative effects of smoking on the outcomes of periodontal therapy Synbiotic were defined as a mixture of probiotics and prebiotics that beneficially affects the host by improving the survival and implantation of live microbial dietary supplements in the gastrointestinal tract, by selectively stimulating the growth and/or by activating the metabolism of one or a limited number of health-promoting bacteria, and thus improving host welfare. Also in some cases, this may lead to a competitive advantage for the probiotics among with other bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects
* Clinical diagnosis of gingivitis

Exclusion Criteria:

* Subjects who had used any systemic antibiotics in the previous 3 months,
* Subjects who had used a product containing probiotics in the previous month
* Systemic disease or condition that could interfere with the study results
* Ongoing drug therapy that could affect the signs of gingivitis
* Subjects who were received periodontal treatment in the last 6 months and
* Allergic to milk and milk products

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2015-06-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Interleukin (IL)-6 level of GCF at 2 months | baseline, 1st and 2nd months
  GCF samples were collected with paper strips and IL-6 levels of GCF were measured using commercial kits by using ELISA method
Change from Baseline IL-8 level of GCF at 2 months | baseline, 1st and 2nd months
  GCF samples were collected with paper strips and IL-8 levels of GCF were measured using commercial kits by using ELISA method
Change from Baseline IL-10 level of GCF at 2 months | baseline, 1st and 2nd months
  GCF samples were collected with paper strips and IL-10 levels of GCF were measured using commercial kits by using ELISA method

SECONDARY OUTCOMES:
Change from Baseline GCF volume at 2 months | baseline, 1st and 2nd months
  Clinical parameter
Change from Baseline Gingival Index at 2 months | baseline, 1st and 2nd months
  Clinical parameter
Change from Baseline Plaque Index at 2 months | baseline, 1st and 2nd months
  Clinical parameter

IPD SHARING:
Plan to Share IPD: Yes
Randomization was performed by one researcher that had never any role in participant's treatment and clinical measurement processes (E.O.E). Patients' all measurements and treatments were made by a single researcher who doesn't know in which group participants were included (N.E.).
Supporting Information: Study Protocol, CSR
Time Frame: study protocol : at the beginning of the study (july 2014) Clinical Study Report (CSR): july 2014, january 2015, july 2015, january 2016, april 2016
Access Criteria: study protocol : with all researchers Clinical Study Report (CSR): Interviewed with all researchers by face to face

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03455192/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03455192/SAP_001.pdf